CLINICAL TRIAL: NCT02351505
Title: An Investigator-Sponsored Phase 2 Study of Single Agent Selinexor (KPT-330) in Patients With Relapsed Small Cell Lung Cancer
Brief Title: Selinexor in Treating Patients With Relapsed Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: Erin Bertino (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Erin Bertino, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14136; NCI-2014-02489 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Recurrent Small Cell Lung Carcinoma
Keywords: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selinexor) (Experimental): Patients receive selinexor PO twice weekly. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selinexor; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial studies how well selinexor work in treating patients with small-cell lung cancer that has returned after a period of improvement. One specific way cancer cells continue to grow is by getting rid of certain proteins called "tumor suppressor proteins: that would normally cause cancer cells to die. Selinexor works by trapping "tumor suppressing proteins" within the cell and may cause the cancer cells to die or stop growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of single agent selinexor as measured by progression free survival (PFS) in patients with relapsed chemotherapy-sensitive small cell lung cancer.

SECONDARY OBJECTIVES:

I. To evaluate the objective tumor response rate and disease control rate as determined by radiographic response.

II. To evaluate the overall survival (OS) in patients with relapsed small cell lung cancer.

III. To evaluate safety and tolerability of single agent selinexor in these patient populations.

IV. Comparison between each patient's time to progression (TTP) on selinexor with the TTP of his/her previous therapy(ies).

V. To evaluate correlative endpoints including tumor biopsy and analysis of secreted factors, leukocyte ribonucleic acid (RNA) analysis.

TERTIARY OBJECTIVES:

I. Analysis of secreted factors (nerve growth factor [NGF], brain-derived neurotrophic factor [BDNF]).

II. Tumor biopsy (baseline and cycle 2).

OUTLINE:

Patients receive selinexor orally (PO) twice weekly. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 3 months, every 3 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines
* Patients should have estimated life expectancy of > 3 months at study entry
* Patients with relapsed small cell lung cancer - diagnosis must be histologically confirmed
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at the time of study entry
* Objective evidence of disease progression on study entry
* Prior systemic anticancer therapy: patients will have received no more than 2 prior chemotherapy regimens; the regimen(s) may have included biological, molecularly targeted or immune therapies; patients with primary refractory disease (i.e., those patients with progressive disease on first line chemotherapy) and patients with disease relapse within 90 days of completion of initial chemotherapy (chemotherapy resistant) are excluded; patients with limited stage small cell lung cancer (SCLC) and systemic relapse who are not felt to be candidates for repeat platinum-based chemotherapy at relapse are eligible for enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) > 1000/mm^3
* Platelet count > 75,000 mm^3
* Total bilirubin < 2 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN)
* Alanine aminotransferase (ALT) < 2.5 times ULN; in the case of known (radiological and/or biopsy documented) liver metastasis, ALT < 5.0 times ULN is acceptable
* Albumin >= 3.0 mg/dl
* Estimated creatinine clearance of >= 30 mL/min, calculated using the formula of Cockroft and Gault
* Amylase =< 1.5 x ULN
* Lipase =< 1.5 x ULN
* Alkaline phosphatase limit =< 2.5 x ULN
* Female patients of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening; male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Resolution to grade =< 1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v4.03) of all clinically significant toxic effects of prior anti-cancer therapy (with the exception neuropathy, which may be =< grade 2 within 14 days prior to cycle 1 day 1)
* Available archival tumor tissue or willingness to undergo repeat biopsy is required at trial initiation

Exclusion Criteria:

* Primary refractory disease (progressive disease on initial platinum based chemotherapy) or chemotherapy-resistant disease (disease progression within 90 days of completion of initial chemotherapy)
* Patients who are pregnant or lactating
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy =< 2 weeks prior to cycle 1 day 1; any clinical trial therapy (including investigational anti-cancer study) =< 3 weeks prior to cycle 1 day 1
* Prior treatment with selinexor
* Major surgery within 3 weeks before day 1
* Unstable cardiovascular function:

  * Electrocardiogram (ECG) abnormalities requiring treatment, or
  * Congestive heart failure (CHF) of New York Heart Association (NYHA) class >= 3
  * Myocardial infarction (MI) within 3 months
  * Symptomatic ischemia or angina
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study
* Known to be human immunodeficiency virus (HIV) seropositive
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) RNA or hepatitis B surface antigen (HBsAg) (hepatitis B virus [HBV] surface antigen)
* Serious psychiatric or medical conditions that could interfere with treatment
* History of seizures, movement disorders or cerebrovascular accident within the past 5 years prior to cycle 1 day 1
* Concurrent therapy with approved or investigational anticancer therapeutic other than steroids
* Patients with > 3 liver metastases at time of enrollment
* Patients with coagulation problems and active bleeding in the last month (peptic ulcer, epistaxis, spontaneous bleeding)
* Patients with significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea or inability to swallow oral medications
* Patients who are severely underweight (body mass index [BMI] less than 17) or patients with a body surface area (BSA) < 1.4 m^2 as calculated per Dubois 1916 or Mosteller 1987
* Uncontrolled brain metastases or leptomeningeal involvement; patients with brain metastases are permitted if they have received appropriate therapy and demonstrated control of the brain metastases or leptomeningeal disease following therapy; patients with known brain metastases will require magnetic resonance imaging (MRI) brain to demonstrate disease control prior to enrollment (lack of symptom progression for two weeks off therapeutic doses of steroids, excluding chronic steroids used for control of chronic obstructive pulmonary disease [COPD])
* Prior cancer diagnosis is allowed if patient is disease-free for >= 3 years, or disease free for < 3 years for treated basal cell/ squamous cell skin cancer or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bertino, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Selinexor (KPT-330): Patients receive selinexor PO twice weekly. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Arm A: Selinexor (KPT-330)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Selinexor (KPT-330): Patients receive selinexor PO twice weekly. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Estimated by the method of Kaplan and Meier for each cohort. Appropriate one-sided 90% confidence boundary will also be calculated for the final test Kaplan-Meyer test statistic at 12 weeks.
Time Frame: Time from the date of study registration to the date of disease progression or to the date of last observation when no event (disease progression) has occurred, assessed up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate (Complete Response [CR] or Partial Response [PR]) by RECIST
Description: The overall response rate will be calculated as the number of PRs and CRs divided by the total number of evaluable patients. Estimates will be accompanied by exact binomial confidence intervals as well.
Time Frame: Up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Control Rate (CR, PR, and Stable Disease)
Description: Estimates will be accompanied by exact binomial confidence intervals.
Time Frame: Up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier curves will be used to estimate overall survival. Consider Cox proportional hazards models to explore a limited set of confounding factors.
Time Frame: Date of study registration to the date of event (i.e., death) or the date of last follow-up if no event has occurred at their last evaluation assessed up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of Adverse Events Defined as Adverse Events That Are Classified as Either Not Related, Possibly, Probably, or Definitely Related to Study Treatment as Per NCI CTCAE v4.0
Description: Summarized by descriptive statistics for each of the disease cohorts. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. In addition, review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing.
Time Frame: Up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Severe (Grade 3+) Adverse Events or Toxicities as Per NCI CTCAE v4.0
Description: The incidence of severe (grade 3+) adverse events or toxicities will be described.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 1
percentage of patients
  Fatigue | 100
  Generalized muscle weakness | 100
  Bilateral Lower Extrem Edema | 100
  Hyperglycemia | 100
  Hyponatremia | 100

7. Secondary Outcome: Tolerability of the Regimen Assessed Through Number of Patients Who Required Dose Modifications and/or Dose Delays
Time Frame: Up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

8. Secondary Outcome: Proportion of Patients Who go Off Treatment Due to Adverse Reactions or Even Those Who Refuse Further Treatment for Lesser Toxicities That Inhibit Their Willingness to Continue Participation on the Trial
Time Frame: Up to 4 years
Population: Unable to analyze data due to only 1 patient being enrolled on the study
Arm/Group | Arm A: Selinexor (KPT-330)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Frequency and severity of adverse events and tolerability of the regimen were collected and summarized by descriptive statistics for each of the disease cohorts. As per NCI CTCAE v4.0, the term toxicity is defined as adverse events that are classified as either not related, possibly, probably, or definitely related to study treatment.
Arm/Group | Arm A: Selinexor (KPT-330)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Selinexor (KPT-330) (N=1)
Activated PTT prolonged (Investigations) | 1 (1) — PTT (Partial Thromboplastin Time)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Depressed level of conciousness (Nervous system disorders) | 1 (1)
Eye disorder-decreased visual acuity (Eye disorders) | 1 (1)
Fall (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — arms and legs
Headache (Nervous system disorders) | 1 (1) — intermittent
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Edema (General disorders) | 1 (1) — Bilateral extremities
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial was closed early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes